CLINICAL TRIAL: NCT05855499
Title: Plasma on Chronic Wounds for Epidermal Regeneration - Randomized, Controlled Clinical Trial to Investigate the Efficacy of Plasma Therapy for the Treatment of Chronic, Non-healing Wounds in Comparison to Standard Wound Therapy -
Brief Title: Plasma on Chronic Wounds for Epidermal Regeneration
Acronym: POWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coldplasmatech (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPT2019_01
Record Dates: First submitted 2023-04-24; First posted 2023-05-11 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Chronic Ulcer of Lower Extremity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma (CAPT) (Experimental): Conventional wound treatment according to S3 guideline, 3 visits weekly for 4 weeks, additive plasma treatment during each visit.
  Interventions: Device: CPtcube, CPTpatch
- Standard wound treatment (SWT) (No Intervention): conventional wound treatment according to S3 guideline, 3 visits weekly for 4 weeks

INTERVENTIONS:
Device: CPtcube, CPTpatch — This study investigates the effectiveness of a system for reproducible application of cold plasma on larger areas and observes the effect of a 4-week additional plasma treatment on wound healing of large chronic wounds.
  Arms: Plasma (CAPT)

SUMMARY:
Every year, 5 million people throughout Germany suffer from extensive, often chronic wounds. Cold plasma is an innovative therapeutic approach in the treatment of these persistent tissue defects. However, previous therapy options with cold plasma are very time-consuming, especially with increasing wound area, and are also strongly dependent on the skill of the practitioner.

This study investigates the effectiveness of a system for reproducible application of cold plasma on larger areas and observes the effect of a 4-week additional plasma treatment on wound healing of large chronic wounds. The patient-related benefit of such an additional treatment will also be evaluated. Both study arms will receive guideline-based wound therapy, which is the current gold standard.

DETAILED DESCRIPTION:
The clinical trial investigates the efficacy of an additional 4-week initial plasma therapy (CAPT) in direct comparison to standard guideline-based wound therapy (SWT) alone. The reactivation of healing of chronic, non-healing wounds will be assessed. This reactivation is primarily measured by the reduction of wound area, a valid and clinically accepted parameter for wound healing. A large number of RCTs and cohort studies demonstrate a strong correlation between the reduction in wound area at 4 weeks and the therapy outcome at 12 and 20 weeks.

In addition to wound area reduction, other clinical parameters such as wound volume, wound closure, percentage of necrotic and fibrotic tissue, percentage of granulation tissue, wound exudate, and microflora are recorded. By recording these secondary endpoints, it is possible to closely track and analyse changes in wound condition induced by cold plasma.

Another focus of the clinical trial is the evaluation of patient-related outcomes such as frequency of occurrence of infections, perception of pain, occurrence of adverse events, frequency of hospitalization, and change in quality of life. These events are fully documented to evaluate the safety of the treatment and to rule out potential risks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are divided into patient-specific and wound-specific criteria.

Patient Criteria:

* Patient must be at least 18 years old (legal age) and legally competent
* The patient has at least one diagnosed chronic (existing for at least 8 weeks), non-healing wound due to a UCA or UCV on the lower leg, below the knee
* There is a signed consent form dated by the patient's own hand

Wound Criteria:

* In case of multiple wounds, the largest wound by area will be included in the study if it meets all inclusion criteria and no exclusion criteria and is suitable for use of the investigational product. The target wound is at least 2 cm away from the other wound(s)
* The wound was diagnosed - at the time of planned inclusion - more than 8 weeks ago and classified as a chronic wound
* The initial wound area is 5 cm²-100 cm2
* The wound can be enclosed completely by the plasma applicator (10 cm x 10 cm)
* The wound is not undermined
* The wound is located on the lower leg

Exclusion Criteria:

The exclusion criteria are divided into patient-specific and wound-specific criteria.

Patient Criteria:

* The patient is younger than 18 years and/or lacks legal capacity
* The patient has already participated in this study
* The patient is already participating in another interventional study
* Pregnant or breastfeeding patients
* The patient has an implanted pacemaker, defibrillator or other active implants
* The patient has a light/sun allergy
* The patient has a silicone allergy
* The patient has had a thrombosis within the last 3 months
* The patient has a systemic and/or chronic infectious disease (e.g., HIV, tuberculosis, hepatitis)
* The patient has a tumour disease
* An ongoing or recently completed chemotherapy or radiotherapy
* The patient is undergoing severe endogenous or drug immunosuppression
* The patient is receiving systemic antibiotic treatment or is receiving/needing antiseptic/antibiotic wound therapy in/near the wound
* The patient does not have the necessary revascularization (paVK)
* The patient requires vital instrumental monitoring in the sense of "basic monitoring": near-patient respiratory gas measurement (oxygen, carbon dioxide and inhalation anaesthetic), pulse oximeter, ECG monitoring, blood pressure measurement (non-invasive), an oscillometric blood pressure measurement with automatic mode
* Existing alcohol or drug abuse
* The patient requires dialysis

Wound Criteria:

* The wound is not a chronic wound as defined by study protocol
* The wound is difficult to access or close to exposed vessels
* The wound is critically colonized or infected
* Acute infections in the wound area (radius 5 cm)
* The wound is bleeding profusely. This does not include bleeding immediately after debridement
* The wound is undermined
* The wound is located at the knee or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in area of chronic wounds | 3 visits weekly for 4 weeks, follow-up at at 12 and 20 weeks
  The clinical trial is based on the following primary null hypothesis (H0):
  There is no significant difference in terms of reduction in area of chronic wounds between standard guideline-based wound therapy with and without initial 4-week plasma treatment.
  The associated alternative hypothesis (HA) is:
  There is a significant difference in terms of reduction in area of chronic wounds between standard guideline-based wound therapy with and without initial 4 weeks of plasma treatment

SECONDARY OUTCOMES:
Wound closures | during the 4-week active treatment phase, after 3 and after 6 months
  Number of patients with wound closures achieved during the 4-week active treatment phase or in the period after the active treatment phase (3 or 6 months after last visit).
Change in wound pain | during the 6-month observation period
  Change in wound pain during activity or at rest during the 6-month observation period. Pain was assessed using an NRS with values ranging from 0 to 10.
Change in quality of life | during the 6-month observation period
  Change in quality of life, assessed using a wound-specific questionnaire (Wound-QoL) and a generic quality-of-life questionnaire (SF-12), at the end of the treatment phase, at wound closure, at early treatment discontinuation, and during the two FU time points, each compared with the start of treatment.
Amount of germs/bacteria in the wound bed | during the 4-week active treatment phase
  For this purpose, swabs are taken before and after treatment. The swabs are then examined in the laboratory with regard to the microflora (germ type and resistance).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Banaschik, Dr., Study Director — Coldplasmatech; Isabel Zänker, Dr., Principal Investigator — Thüringen-Kliniken
Locations (8):
- Germany (8):
  - Universitäts-Hautklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Zentrum Rothenaicher, München, Bavaria
  - Zentrum Regensburg, Regensburg, Bavaria
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Katholisches Klinikum Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
  - Verbund Thüringen-Kliniken "Georgius Agricola", Saalfeld, Thuringia

IPD SHARING:
Plan to Share IPD: Undecided